CLINICAL TRIAL: NCT00680771
Title: The Psychoneuroimmunology of Insomnia: Response to a Vaccine Challenge
Brief Title: The Psychoneuroimmunology of Insomnia
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Wilfred Pigeon, Assistant Professor of Psychiatry, University of Rochester
Other Study IDs: RSRB # 19132; 1K23NR010408 (NIH)
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Results first posted 2012-10-17 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-09

CONDITIONS: Primary Insomnia
Keywords: Primary Insomnia; Insomnia; Good Sleepers; Hep B; Vaccine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Primary Insomnia
- 2: Good Sleepers

SUMMARY:
Chronic insomnia affects approximately 8-9% of the population. The prevalence of this disorder rises dramatically across the lifespan, especially so in women. When it is chronic, insomnia is associated with increased fatigue, cognitive impairment, mood disturbance, physical complaints, diminished quality of life and increased health care consumption. There is also more limited evidence (based on epidemiologic studies or experimental studies in healthy subjects) that insomnia and/or sleep loss may be a risk factor for hypertension and/or cardiovascular disease and increased mortality.

Despite its prevalence and consequences, the pathophysiology of insomnia and, specifically, the pathway by which morbidity risk is conferred, has been relatively unstudied. With respect to medical illness in particular, insomnia may confer risk in several ways, including: 1) an inherent compromise in the restorative/conservative function of sleep, 2) the deleterious effects of "hyperarousal" and/or HPA axis abnormalities on end organ integrity and function, and/or 3) diminished immunocompetence. This study focuses on the last of these possibilities, the relationship between immune function and sleep.

The study compares immune response to a vaccine challenge in two groups: good sleepers and patients with chronic insomnia. The primary study hypothesis is that the insomnia group will have a decreased rate of adaptive immune response to the vaccine challenge than that of the good sleeper group.

ELIGIBILITY:
Inclusion Criteria:

Their sleep schedule will include a typical bedtime of between 9:00 p.m. and 12:00 a.m. to minimize circadian rhythm influences on the diagnoses of Primary Insomnia (PI).

PIs will also meet the sleep disturbance criteria of the Pittsburgh Sleep Quality Index(PSQI) > 5 and the Insomnia Severity Index (ISI)> 15 and one of the following minimal characteristics both at intake and as an average profile from the two weeks of baseline diaries: > 30 min. sleep-onset latency (SL), > 30 min. of wake after sleep-onset (WASO), Early Morning Awakening >30 min. prior to the desired wake up time, or any two of the above complaints (Mixed Insomnia); Total Sleep Time (TST) < 6 hours [unless the Sleep Efficiency is < 80%] and the problem frequency must be > 3 nights/week; problem duration > 6 months.

Good Sleeper participants will report that they obtain enough sleep and that their sleep is restorative with average SL and WASO < 15 minutes, TST > 6 hours ESS < 5 on the ESS, < 5 on the PSQI, and < 7 on the ISI.

Exclusion Criteria for All Subjects

* any conditions contraindicated by the vaccine manufacturer or any history of allergic reactions to vaccines
* Undergoing and/or taking immunosuppressive therapies
* Sero-positive for Hep B antibodies
* Inadequate language comprehension
* Menopause, peri-menopause or premenstrual syndrome
* Pregnancy
* Unstable medical or psychiatric illness
* History of head injury with a sustained loss of consciousness
* Evidence of active illicit substance use or fitting criteria for alcohol abuse or dependence
* Use of medications thought to alter sleep such as stimulants, sedating antidepressants, and hypnotics
* Symptoms suggestive of sleep disorders other than Insomnia
* Polysomnographic data indicating sleep disorders other than Insomnia

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred R Pigeon, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Sleep Research Laboratory, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre-menopausal women aged 25-50 with either Primary Insomnia (PI) or Good Sleep (GS) were recruited from posters, flyers, and newspaper advertisements in the Rochester, NY region during the period of 2008-2010.
Pre-assignment Details: There were two study groups, but this did not involve random assignment. Group assignment to either Primary Insomnia or Good Sleeper was based on subjective (sleep diaries and validated instruments)and objective (polysomnography) measures of sleep. Twenty-eight subjects were enrolled.
Groups:
- Primary Insomnia: Subjects meeting criteria for primary insomnia.
- Good Sleepers: Subjects meeting criteira for Good Sleepers
Period: Overall Study
Arm/Group | Primary Insomnia | Good Sleepers
Started | 15 | 13
Completed | 9 | 11
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Sleep Apnea suspected after PSG | 1 | 0
Not completed — Prior Exposure to Hepatitus B Vaccine | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Primary Insomnia: patients meeting criteria for primary insomnia.
- Good Sleepers: participants meetoing criteira for Good Sleepers
- Total: Total of all reporting groups
Arm/Group | Primary Insomnia | Good Sleepers | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Positive Antibody Response
Description: Sero-Response to the Hepatitis B vaccine, defined as reaching or exceeding a Hepatitis B surface antigen level of greater than or equal to 10mIU/mL.
Time Frame: 3 Months after initial vaccination
Population: From subjects with complete data only.
Measure: Number; unit: participants
Arm/Group | Primary Insomnia | Good Sleepers
Number analyzed (Participants) | 8 | 11
participants | 7 | 7

ADVERSE EVENTS:
Arm/Group | Primary Insomnia | Good Sleepers
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13

LIMITATIONS AND CAVEATS:
Sample size limited by much higher than expected number of otherwise eligible participants having alrady been exposed to Hep B vaccine or virus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No